CLINICAL TRIAL: NCT03590834
Title: Obesity Prevention in Head Start: Míranos! Program
Brief Title: Míranos! Program, a Preschool Obesity Prevention RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at San Antonio (Other)
Collaborators: University of Texas at Austin (Other); University of Maryland (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Family Service Association of San Antonio Inc. (Unknown); Parent/Child Incorporated (PCI) of San Antonio and Bexar County (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DK109323 (NIH); R01DK109323 (NIH)
Record Dates: First submitted 2018-06-27; First posted 2018-07-18 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Healthy Eating; Physical Activity; Health Knowledge, Attitudes, Practice; Gross Motor Development
MeSH Terms: conditions — Obesity; Motor Activity; Behavior

STUDY DESIGN:
Masking Description: The parents of the children were informed that their Head Start center will be randomly assigned to one of the three study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Center-based intervention (Experimental): In-person, child-focused intervention taking place only at the Head Start centers
  Interventions: Behavioral: Center-based Intervention
- Center-and-home-based intervention (Experimental): In-person, child-focused intervention taking place only at the Head Start centers. Delivered in-person at Head Start centers and the family home.
  Interventions: Behavioral: Home-based Intervention
- Active Control (Active Comparator): Active comparison group
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Center-based Intervention — 1. Center nutrition and physical activity policy modification to increase fruit and vegetable servings and more physical activity throughout the day
  2. Staff training and technical assistance
  3. Health education on healthy habits (diet, physical activity, sleep, screen time) using the Sesame Workshop Healthy Habits for Life (HHL) resource kit
  4. Health contests
  5. Gross motor and physical activity program
  6. Miranos! activity cards based on children storybooks
  Other Names: CBI
  Arms: Center-based intervention
Behavioral: Home-based Intervention — 1. Monthly interactive poster education sessions led by parent peer educators during child pick-up time. Held at Head Start Center. These sessions include family health challenges and take-home activities.
  2. Three Home Visits delivered by Head Start staff. Obesity prevention goal-setting integrated into existing Head Start home visits
  3. 16 semi-monthly, Family Newsletters with stories, tips, and strategies to promote healthy habits for preschool children
  4. Incorporating activities related to PA, nutrition and sleep into existing Head Start Center Summer Calendars
  Other Names: C+HBI
  Arms: Center-and-home-based intervention
Behavioral: Active Control — Children will receive Head-Start-approved health education program for children: "I Am Moving, I Am Learning". In addition, the investigators will deliver an early childhood literacy program to all active control children to increase buy-in and retention.
  Arms: Active Control

SUMMARY:
The prevalence of obesity remains high in American children aged 2-5 while one in three Head Start children is overweight or obese. The proposed study is designed to test the efficacy of an early childhood obesity prevention program which promotes healthy growth in predominantly Latino children in Head Start.

The program is a group clustered randomized controlled trial in partnership with two local Head Start organizations to address key enablers and barriers in obesity prevention in young children. The study has three specific aims:

1. To test the efficacy of the Miranos! intervention on healthy weight growth (primary outcome) in normal weight, overweight, and obese children.
2. To test the impact of the Miranos! intervention on children's physical activity, sedentary behavior, sleep, and dietary behaviors (secondary outcomes).
3. To evaluate cost-effectiveness of the Miranos! intervention.

Miranos! will be delivered in Fall and Spring (8 months) and followed by a summer health campaign.

DETAILED DESCRIPTION:
Using a three-arm design, 12 Head Start (HS) centers in equal number will be randomly assigned to one of three conditions: 1) a combined center- and home-based intervention, 2) center-based intervention only, or 3) active control. The interventions will be delivered during the academic year (an 8-month [mo] period). A total of 525 3-year-old children (52% females; in two cohorts) will be enrolled in the study at baseline and followed prospectively one-year post-intervention. The first cohort will be recruited in summer 2018. The second cohort will be recruited in summer 2019.

Data collection will be conducted at baseline (T0), immediate post-intervention (T1), and 1-year post-intervention follow-up (T2) and include children's height, weight, accelerometry-based PA and sedentary behavior, TV watching and sleep by parent reports, gross motor development, dietary intakes, food preference. Information on family background, parental PA- and nutrition-related practices, parental weight and health behaviors, PA and nutrition policies and environments at the center and home, and costs associated with intervention delivery will be collected. The primary endpoint for the study is the BMI at the posttest immediately following the completion of the intervention (T1).

Recruitment: Participant recruitment will take place during summer by sending a recruitment packet to child's home. This packet includes: study information sheet, recruitment flyer, informed consent form, a letter from center director and study PIs.

Process Evaluation: The process evaluation is informed by the NIH Behavior Change Consortium Treatment Fidelity Workgroup's best practice recommendations and recent multi-component RCTs. Míranos! has multiple components with multiple activities, the investigators will use many indicators to evaluate the fidelity and completeness of the implementation of all components and determine contribution of each component by linking it to the primary and secondary outcomes. The investigators will collect both quantitative/qualitative data to assess cross-site treatment consistency, non-treatment-related effects, and document protocol changes.

First, intervention dose delivered will be measured by: 1) pre-/post-study center environmental assessment by the Environment and Policy Assessment and Observations (EPAO) and auditing of meal menus; 2) completion of delivery schedule of staff, peer leader training, parent education sessions, home visits; 3) evaluation of staff, peer leader training; 4) monthly auditing of weekly lesson plans; and 5) monthly checklist of use of Míranos! Activity Cards, children's story books, HHL learning activities.

Second, the intervention dose received will be assessed by: 1) attendance records of staff, peer leader training, parent education sessions; 2) certification test of staff, peer leader training; 3) monthly staff evaluation (rating scale) of children's learning of HHL content, gross motor skills, eating behaviors; 4) post-study parent intercept interviews; and 5) post-study focus groups on program delivery process with staff (n=24) and parents (n=32).

Third, participants' responses to the intervention will be evaluated by: 1) random observations of staff behavior (rating scale) during outdoor play and lunch by research staff; 2) assessments on children's PA by the System for Observing Fitness Instruction Time for Preschoolers and diet by group plate waste test in 3 randomly selected centers; 3) in-depth interviews with staff (n=48) for program feedback; and 4) post-study staff and parent evaluation (rating scale) of satisfaction with intervention components/activities.

ELIGIBILITY:
Inclusion Criteria:

* The child must be enrolled in a full-day Head Start center
* The child must be 3 years old at baseline, one child per family, parental consent

Exclusion Criteria:

* N/A

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 525 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Baseline, 8 months, 21 months
  Child's height and weight will be measured twice with no shoes and light clothing in an area separated by a privacy screen, using a stadiometer and digital weight scale. Discrepancy between the two measures must be ≤0.2 cm and≤ 0.10 kg. BMI, BMI-percentile, and zBMI for age and gender will be calculated using the average of the two measures based CDC Growth Charts.

SECONDARY OUTCOMES:
Change in Physical Activity, Sedentary Activity, and Sleep | Baseline, 8 months, 21 months
  7-d accelerometry to measure the minutes of light-, moderate- and vigorous-intensity physical activity, sedentary activity, and sleep/day
Change in Parent report of screen time and sleep | Baseline, 8 months, 21 months
  7-d parent log to track time that child spends watching TV/DVD and sleeping each day
Change in Fruit, vegetable, and beverage consumption | Baseline, 8 months, 21 months
  Assessment of children's consumption of fruits, vegetables and beverages by screener on the frequency and portion size of food items that will be completed by the parents as well as aggregate plate waste to asses intake at sites.
Change in Food preference | Baseline, 8 months, 21 months
  A computer-assisted pictorial test to measure young children's preferences for healthy food
Change in Parent Behavior | Baseline, 8 months, 21 months
  Parents will complete: 1) the Home Health Environment survey, 2) the Parenting Strategies for Eating and Activity Scale, 3) health knowledge assessment; and 4) parental confidence/self-efficacy scale.
Demographic Information | Baseline
  Information will be collected from the parents on family socioeconomic status (parent education, income, employment, health insurance, food insecurity, race/ethnicity, age, sex), acculturation (a 12-item bidirectional measure), family structure, type of residence, and family health history at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Zenong Yin, PhD, Principal Investigator — University of Texas at San Antonio; Deborah Parra-Medina, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after data has been analyzed for primary and secondary outcome measures
Access Criteria: Data will be made available for research educational purposes.

REFERENCES:
- [Background] Yin Z, Ullevig SL, Sosa E, Liang Y, Olmstead T, Howard JT, Errisuriz VL, Estrada VM, Martinez CE, He M, Small S, Schoenmakers C, Parra-Medina D. Study protocol for a cluster randomized controlled trial to test " inverted exclamation markMiranos! Look at Us, We Are Healthy!" - an early childhood obesity prevention program. BMC Pediatr. 2019 Jun 10;19(1):190. doi: 10.1186/s12887-019-1541-4. PMID 31179916
- [Background] Ullevig SL, Parra-Medina D, Liang Y, Howard J, Sosa E, Estrada-Coats VM, Errisuriz V, Li S, Yin Z. Impact of inverted exclamation markMiranos! on parent-reported home-based healthy energy balance-related behaviors in low-income Latino preschool children: a clustered randomized controlled trial. Int J Behav Nutr Phys Act. 2023 Mar 21;20(1):33. doi: 10.1186/s12966-023-01427-z. PMID 36944986
- [Background] Yin Z, Liang Y, Howard JT, Errisuriz V, Estrada VM, Martinez C, Li S, Ullevig SL, Sosa E, Olmstead T, Small S, Ward DS, Parra-Medina D. inverted exclamation markMiranos! a comprehensive preschool obesity prevention programme in low-income Latino children: 1-year results of a clustered randomised controlled trial. Public Health Nutr. 2023 Feb;26(2):476-487. doi: 10.1017/S1368980022002439. Epub 2022 Nov 11. PMID 36357340